CLINICAL TRIAL: NCT05065957
Title: Open-Label, Multicenter, Phase II/III Study of Combination Therapy of D07001-Softgel Capsules and Xeloda/TS-1 in Subjects With Advanced Biliary Tract Cancer After Gemcitabine and Cisplatin-Based Treatment Failure
Brief Title: Study of Combination Therapy of D07001-Softgel Capsules and Xeloda/TS-1 in Subjects With Advanced Biliary Tract Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: InnoPharmax Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Inno-GO-05
Record Dates: First submitted 2021-09-07; First posted 2021-10-04 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Capecitabine; titanium silicide; Control Groups

STUDY DESIGN:
Intervention Model Description: In phase IIa, a modified 3+3 dose-finding design trial will be conducted to identify the selected dose of the combination of D07001-softgel capsules plus Xeloda (or TS-1). After the dose-finding stage will be completed, a phase IIb/III adaptive design, open label, multicenter, active controlled, parallel-group trial will be implemented and incorporated into a dose-expansion stage to evaluate the efficacy and safety of D07001-softgel capsules plus Xeloda.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase IIa:Dose-Finding Stage (Experimental): Level -5: 20 mg D07001-softgel capsules plus 625 mg/m^2 Xeloda (or 20/30/40 mg TS-1).
  Level -4: 40 mg D07001-softgel capsules plus 625 mg/m^2 Xeloda (or 20/30/40 mg TS-1).
  Level -3: 60 mg D07001-softgel capsules plus 625 mg/m^2 Xeloda (or 20/30/40 mg TS-1).
  Level -2: 80 mg D07001-softgel capsules plus 625 mg/m^2 Xeloda (or 20/30/40 mg TS-1).
  Level -1 (starting dose): 100 mg D07001-softgel capsules plus 625 mg/m^2 Xeloda (or 20/30/40 mg TS-1).
  Level 1: 100 mg D07001-softgel capsules plus 800 mg/m^2 Xeloda (or 30/40/50 mg TS-1).
  Level 2: 100 mg D07001-softgel capsules plus 1000 mg/m^2 Xeloda (or 40/50/60 mg TS-1).
  Interventions: Drug: D07001-softgel capsules + Xeloda (or TS-1)
- Phase IIb/III: Dose Expansion Stage (Active Comparator): ASC+ D07001-softgel capsules plus Xeloda (or TS-1)
  ASC+mFOLFOX (5-FU+Oxalipatin+folinic acid)
  Interventions: Drug: D07001-softgel capsules + Xeloda (or TS-1); Drug: mFOLFOX

INTERVENTIONS:
Drug: D07001-softgel capsules + Xeloda (or TS-1) — D07001-softgel capsules: 3 times per week (on Days 1, 3, 5, 8, 10, 12, 15, 17, and 19 of a 21-day cycle, 9 doses per cycle).
  Xeloda (or TS-1): twice daily for 14 consecutive days followed by 7 days rest (1 treatment cycle)
  Other Names: Treatment group
Drug: mFOLFOX — intravenous infusion on Day 1 for 14-day cycle
  Other Names: Control group
  Arms: Phase IIb/III: Dose Expansion Stage

SUMMARY:
The primary objective are:

To assess the safety and tolerability of the combination of D07001-softgel capsules and Xeloda/TS-1.

To evaluate the efficacy of the combination of D07001-softgel capsules and Xeloda/TS-1, as assessed by disease control rate (DCR).

DETAILED DESCRIPTION:
This open label, multicenter study will be conducted in 2 stages: a dose-finding stage (Phase IIa) and a dose-expansion stage (Phase IIb/III).

In phase IIa, eligible patients will be assigned to receive oral D07001-softgel on Days 1, 3, 5, 8, 10, 12, 15, 17, and 19 of a 21-day cycle (9 doses per cycle) and Xeloda (or TS-1) twice daily on Day 1-14 of a 21-day cycle.

A modified 3+3 dose-finding design method will be applied to identify dose-limiting toxicities (DLTs) and establish the selected dose of D07001-softgel capsules plus Xeloda (or TS-1).

In phase IIb/III,the first 40 subjects (20 subjects per arm) will be randomly allocated in a 1:1 ratio in two arms. Arm A will receive active symptom control (ASC) with the selected dose from dose-finding stage of D07001-softgel capsules and Xeloda (or TS-1), in 21-day cycles. In arm B, subjects will receive ASC with mFOLFOX treatment. After the last subject of first 40 subjects will be completed the visit in the end of treatment, an adaptive interim analysis will be planned to re-estimate the required sample size based on the result of DCR if needed. The sponsor team will determine whether the study will be continued or stopped for futility.

If the study continues to proceed, the total subject number will be based on the decision from the results of interim study. The rest of subjects will be randomized to receive the combination of study drug or active-control drug with the same allocation in two arms. Both groups will continue the therapy until disease progression, withdrawn consent, or when another treatment discontinuation criterion is met.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years or older at screening (aged 20 years or older in Taiwan)
2. Histopathological or cytologic diagnosis of unresectable metastatic or locally advanced BTC (cholangiocarcinoma, gallbladder cancer or ampullary carcinoma)
3. Subject must have failed from first line gemcitabine and cisplatin-based chemotherapy
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-1
5. Life expectancy is >12 weeks
6. Adequate bone marrow function, demonstrated by:

   1. Absolute neutrophil count (ANC) ≥1,500 cell/mm3
   2. Platelet count ≥ 100,000 cells/mm3
   3. Hemoglobin ≥ 9 g/dL
7. Adequate liver function, demonstrated by:

   1. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 x upper limit of normal (ULN), or ≤5.0 x ULN in the case of liver metastases
   2. Total bilirubin ≤1.5 x ULN
   3. Albumin ≥3.0 g/dL
   4. International normalized ratio (INR) <1.5
8. Adequate renal function, demonstrated by:

   1. Serum creatinine ≤1.5 x ULN
   2. Creatinine clearance ≥ 50mL/min calculated by Cockcroft-Gault formula or eGFR ≥ 50mL/min/1.73m2 by 2021 CKD-EPI Creatinine Equation
9. A negative serum pregnancy test at screening and is not breastfeeding in woman of childbearing potential
10. Women of childbearing potential or male subjects must use a medically acceptable form of contraception as 2 barrier methods (e.g., combination of condom, diaphragm, or intrauterine device), hormonal contraception (estrogen or progesterone agents) or 1 barrier method in combination with spermicide. Birth control is required 1 month prior to screening, for the duration of their study participation, and for 1 month after the end of the study; female partners of male subjects must adhere to the same birth control methods.
11. Provision of a signed and dated written Informed Consent Form (ICF) prior to any study specific procedures
12. Subject is willing to comply with protocol-required visit schedule and visit requirements
13. No more than 60 days have elapsed between completion of the prior line of chemotherapy or CCRT and enrollment
14. Subject has not received other chemotherapy since first-line treatment

Exclusion Criteria:

1. Have prior chemotherapy regimen other than first line gemcitabine and cisplatin-based therapy for unresectable metastatic or locally advanced BTC Note: prior fluoropyrimidine base (including capecitabine, carmofur (HCFU), doxifluridine, fluorouracil (5-FU), and tegafur) chemotherapy (including fluoropyrimidine monotherapy or combination therapy) are allowed as postsurgical adjuvant therapy.
2. Diagnosis of active malignancy other than BTC within the past 2 years, except nonmelanoma skin carcinoma and carcinoma-in-situ of uterine cervix treated with curative intent
3. Prior discontinuation of gemcitabine because of pulmonary or hepatic toxicity or hemolytic uremic syndrome (HUS) or hypersensitivity, allergic reaction, or intolerance
4. Known or suspected hypersensitivity to capecitabine, tegafur, gimeracil, oteracil potassium, oxaliplatin or other platinum compounds, leucovorin products, folic acid or folinic acid, 5-fluorouracil or their excipients.
5. Prior discontinuation of fluoropyrimidine because of any unexpected or severe reaction.
6. Treatment with brivudine, sorivudine, or its chemically-related analogs ≤ 28 days prior to the date of enrollment.
7. Under flucytosine treatment.
8. Residual toxicity from prior chemotherapy or CCRT that is Grade ≥2 (residual Grade 2 neuropathy and alopecia are permitted)
9. Any GI disorder which would significantly impede absorption of an oral agent
10. Known brain or leptomeningeal metastases
11. Major surgery or definitive ablation-intent (excluding palliative radiotherapy for bone metastasis) radiation therapy within the past 28 days
12. Any active disease or condition that would not permit compliance with the protocol
13. Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, unstable angina, congestive heart failure, or New York Heart Association [NYHA] Grade 2 or greater), or uncontrolled serious cardiac arrhythmia
14. Have documented cerebrovascular disease. Subjects with the disease may be excluded, but if the investigator assesses that they are asymptomatic or well controlled could be enrolled.
15. Have a seizure disorder not controlled on medication (based on decision of Investigator)
16. Received an investigational agent within 28 days of enrollment
17. Have an uncontrolled active viral, bacterial, or systemic fungal infection
18. Known human immunodeficiency virus (HIV) infection
19. Have HBsAg (hepatitis B surface antigen) positive with HBV-DNA ≥2000 copies/ml and/or anti-HCV antibody (HCV) positive with HCV-RNA positive.
20. Received yellow fever vaccine or other live attenuated vaccine(s) within the 4 weeks prior to screening
21. History of drug or alcohol abuse within last year
22. Have any other serious medical condition that, in the Investigator's medical opinion, would preclude safe participation in, and compliance with, a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs)/ serious adverse event (SAEs) | From date of informed consent to 30-day follow-up visit for each subject
  AEs will be assessed via the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
To assess disease control rate (DCR) | From date of randomization until the date of first documented progression, date of death from any cause, or date of withdraw the study for each subject, whichever came first, assessed up to 24 months
  To assess DCR, the percentage of treatment patients who achieved CR, PR, or SD.

SECONDARY OUTCOMES:
Phase IIa and IIb: Pharmacokinetics (PK) of gemcitabine (dFdC), difluorodeoxyuridine (dFdU), capecitabine, 5-FU, Tegafur, Gimeracil, and Oteracil potassium | Cycle 1 Days 1, 8, and 12 (each cycle is 21 days)
  PK parameters (Peak Plasma Concentration (Cmax)) of gemcitabine and Xeloda or TS-1 will be evaluated
Quality of life (QOL) will be assessed using the EORTC questionnaires | Cycle 1 Days 1, and date of withdraw the study (assessed up to 24 months) for each subject (each cycle is 21 days)
  To access healthrelated quality of life of cancer patients participating in clinical trial.
To assess Progression-free survival (PFS) | From date of randomization until the date of first documented progression, date of death from any cause, or date of withdraw the study for each subject, whichever came first, assessed up to 24 months
  To assess PFS, the time from treatment assignment/randomization until objective tumor progression or death
To assess Objective response rate (ORR) | From date of randomization until the date of first documented progression, date of death from any cause, or date of withdraw the study for each subject, whichever came first, assessed up to 24 months
  To assess ORR, the proportion of treated patients who achieved a BOR of CR or PR.
To assess overall survival (OS) | The survival follow-ups will follow every 6 weeks from date of discontinued study drug for up to 24 months till the death of the subject or closure of the study.
  To assess OS, the time from treatment assignment/randomization until death from any case

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, Ph.D, Principal Investigator — National Institute of Cancer Research
Locations (5):
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Cancer Center, Taipei
  - National Taiwan University Hospotal, Taipei
  - Taipei Veterans General Hospital, Taipei